CLINICAL TRIAL: NCT01496768
Title: Effects of Chronic Leucine Supplemetion on Glucose Homeostasis, Body Compositin, Muscle Mass and Strength of Healthy and Young Subjects: a Randomized, Double-blind, and Placebo Controlled Trial
Brief Title: Effects of Chronic Leucine Supplemetion on Glucose Homeostasis, Body Compositin, Muscle Mass and Strength of Healthy and Young Subjects
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Humberto Nicastro, PhD Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20120412
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Effect of Chronic Leucine Supplementation on Glucose Homeostasis, Lipid Profile, Body Composition, and Muscle Mass and Strenght
MeSH Terms: interventions — Leucine; Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Leucine (Experimental)
  Interventions: Dietary Supplement: Leucine
- Alanine (Placebo Comparator)
  Interventions: Dietary Supplement: Alanine

INTERVENTIONS:
Dietary Supplement: Leucine — 7,2 g/day during 3 months
  Arms: Leucine
Dietary Supplement: Alanine — 7,2 g/day during 3 months
  Arms: Alanine

SUMMARY:
This study aims to evaluate the effects of chronic leucine supplemetion on glucose homeostasis, body compositin, muscle mass and strength of healthy and young subjects

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers;
* Healthy;
* Non-users of dietary supplements and drugs
* Not engaged in any regular physical activity program

Exclusion Criteria:

* Vegetarians

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Muscle strenght | 3 months
Body composition | 3 months
Muscle cross-sectional area | 3 months

SECONDARY OUTCOMES:
Glucose homeostasis | 3 months
Lipid profile | 3 months
Systemic inflammation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerolyn de Souza Valente, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo - School of Physical Education and Sports, São Paulo, São Paulo, Brazil